CLINICAL TRIAL: NCT02196649
Title: Prophylactic and Endoscopic Clip Placement to Prevent Clinically Significant Post Wide Field Endoscopic Mucosal Resection Bleeding - a Randomised Controlled Trial.
Brief Title: Clip Placement Following Endoscopic Mucosal Resection - Randomised Trial
Acronym: CuRB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HREC2014/5/4.2(3971)
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic Clipping (Experimental): Participants randomised to the arm will receive endoscopic clips to their defect following EMR.
  Interventions: Device: Endoscopic Clip
- No Endoscopic Clipping (No Intervention): These participants will receive standard of care practice only.

INTERVENTIONS:
Device: Endoscopic Clip
  Arms: Endoscopic Clipping

SUMMARY:
Patients will be randomised to have endoscopic clips applied to the Endoscopic Mucosal Resection (EMR) site following complete removal of the lesion, or will not receive clips and proceed with standard of care.

DETAILED DESCRIPTION:
The outlined literature suggests that colonic post EMR bleeding may be prevented by the use of prophylactic endoscopic clips. There has thus far been no prospective study to confirm this concept. The ideal way to prove the hypothesis is to conduct a randomised controlled trial to evaluated the use of prophylactic clip placement on the EMR resection defect, for the purpose of preventing delayed bleeding in colonic wide field EMR (lesions>20mm). Given the significantly increased rate of bleeding in the proximal colon, clip placement in this location may have the greatest benefit. If it is proven that such a prophylactic technique is effective and safe, it may lead to significantly decreased patient morbidity and health care resources associated with the management delayed bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Can give informed consent to trial participation
* Lesion size greater than 20 mm
* Lesion proximal to and inclusive of mid transverse colon
* Laterally spreading or sessile polyp morphology

Exclusion Criteria:

* Previous resection or attempted resection of lesion
* Clip deployed prior to the completion of the EMR
* Major intraprocedural bleeding not treatable by coagulation
* Endoscopic appearance of invasive malignancy
* Age less than 18 years
* Pregnancy
* Active Inflammatory colonic conditions (e.g. inflammatory bowel disease)
* Use of anticoagulant or antiplatelet agents other than aspirin less than 5 days prior to procedure
* American Society of Anesthesiology (ASA) Grade IV-V

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-10; Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Post-Procedural Bleeding | 14 days
  Clinically significant post colonic wide-field EMR bleeding (CSPEB)

SECONDARY OUTCOMES:
Safety success | 18 months
  Safety - admission rates, adverse outcomes, deaths Rate of initial technical success Duration of procedure Recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Gupta S, Sidhu M, Shahidi N, Vosko S, McKay O, Bahin FF, Zahid S, Whitfield A, Byth K, Brown G, Lee EYT, Williams SJ, Burgess NG, Bourke MJ. Effect of prophylactic endoscopic clip placement on clinically significant post-endoscopic mucosal resection bleeding in the right colon: a single-centre, randomised controlled trial. Lancet Gastroenterol Hepatol. 2022 Feb;7(2):152-160. doi: 10.1016/S2468-1253(21)00384-8. Epub 2021 Nov 18. PMID 34801133